CLINICAL TRIAL: NCT04610593
Title: Effects of a Mindfulness-based Intervention in the Reduction of Stressors, Pain Profile and Quality of Life of People With Chronic Renal Disease in Hemodialysis
Brief Title: Effects of a Mindfulness-based Intervention in Stress, Pain and Quality of Life in People Undergoing Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0017
Record Dates: First submitted 2020-10-09; First posted 2020-10-30 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Renal Insufficiency, Chronic; Kidney Failure, Chronic; Kidney Diseases; Kidney Insufficiency, Chronic; Chronic Kidney Diseases; End-Stage Kidney Disease
Keywords: End-Stage Kidney Disease; Chronic Kidney Diseases; Renal Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will receive a Mindfulness-based intervention for 8 weeks, and after the intervention this participants will continuous their treatment as usual
  Interventions: Behavioral: Mindfulness-based Intervention
- Treatment as Usual (No Intervention): Patients in the control group received treatment as usual in the hemodialysis setting: Carry out hemodialysis sessions three times a week, on alternate days, for approximately 4 hours added to appointments and procedures performed by professionals from different areas (medicine, nursing, nutrition, physical education, social work, pharmacy, psychology).

INTERVENTIONS:
Behavioral: Mindfulness-based Intervention — A mindfulness-based intervention will be developed for chronic hemodialysis patients to be performed during hemotherapy sessions. This is an integrative mind-body program, which is based on the MBRP (Bowen et al., 2014) and BMT (T. Russell, 2015) protocols. The program will be conducted in eight weeks, with a weekly individual session of up to 60 minutes facilitated by an instructor, at the bedside during the HD session. The program aims to develop awareness of bodily sensations, emotions and thoughts, with an attitude of openness, curiosity, kindness and non-judgment. During the sessions will be worked four main techniques of mindfulness meditation: mindfulness in breathing, body scanning, conscious movements and practice of compassion. Participants are invited and encouraged to practice Mindfulness using audios made available during the other HD sessions they undergo during the week, in addition to daily home practice.
  Arms: Intervention Group

SUMMARY:
This project has as main objective to evaluate the effects of a Mindfulness-based intervention (MBI) in the reduction of stressors, pain and quality of life of people with chronic kidney disease undergoing hemodialysis (HD). The investigators hypothesize that this program offered during hemodialysis sessions may modify the pain profile, stressors levels and may improve the quality of life by the people in hemodialysis. This is an incipient field of research at the international level and almost nonexistent in Brazil. Evidence indicates the need for MBIs to be performed during HD sessions, adapted to the context, to facilitate patient compliance, contribute to the management of the discomfort generated during HD and promote health.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is considered a global public health problem, which affects approximately 10% of the world population. Due to partial or total loss of kidney function, the patient needs renal replacement therapy, with hemodialysis (HD) being the therapy most used, having a prevalence of up to 93.1% in Brazil. The restrictions imposed by CKD and the treatment of prolonged HD negatively affect health, increasing stress and decreasing the quality of life (QoL). The restrictions imposed by CKD and the treatment of prolonged HD negatively affect health, increasing stress and decreasing the QoL. Hemodialysis supports life and relieves a series of symptoms; however, it imposes many limitations. Social, financial and family stressors are numerous when dealing with the symptoms of the disease, restrictions and treatment prescriptions. Research shows positive results from Mindfulness-Based Interventions (MBIs) in reducing symptoms of different chronic diseases and mental and physical disorders such as: depression, anxiety, hypertension, cancer, chronic pain, cardiovascular diseases, insomnia, addictive behaviors, and kidney disease, and in improving medication adherence. This is an incipient field of research at the international level and almost nonexistent in Brazil. Evidence indicates the need for MBIs to be performed during HD sessions, adapted to the context, to facilitate patient compliance, contribute to the management of the discomfort generated during HD and promote health. This project has as main objectives to develop and evaluate the effects of a mindfulness-based intervention in the reduction of stressors, pain and quality of life of people undergoing hemodialysis. For this purpose, a randomized controlled pragmatic study with random allocation and blinding of the outcome evaluator will be performed, using quantitative and qualitative measures evaluated within 6 months after the intervention. The results of this research could form a consistent basis for a new and promising field of research that could contribute to improving the health of people undergoing hemodialysis and other populations that need long-term hospital care.

ELIGIBILITY:
Inclusion Criteria:

* Higher than 18 years old;
* Undergoing hemodialysis for at least three months;
* Auditory acuity to listen to Mindfulness practices;
* Be interested in the objectives of this study and be randomized in one of the two groups (MBI or TAU).

Exclusion Criteria:

* Severe cognitive impairment or severe psychiatric disorder diagnosed by the medical staff of the nephrology unit;
* Suicidal ideation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Pain Acceptance | Change from Baseline in AAQ-II at 6 months
  The Acceptance & Action Questionnaire (AAQ-II) is a self-report questionnaire of seven items and aims to measure experiential avoidance. The answers are arranged on a seven-point Likert scale, in which 1 corresponds to "never true" and 7 to "always true". The final scores range from 10 to 70 points, with low scores corresponding to greater acceptance and ability to act in the presence of difficult thinking and emotions.

SECONDARY OUTCOMES:
Renal disease and quality of life | Change from Baseline in KDQOL-SF at 6 months
  The Kidney Disease Quality of Life - Short Form (KDQOL-SF) is a self-reported measure that assesses the functioning and wellbeing of people with kidney disease and on dialysis. This scale is divided in 4 domains: Your Health, Kidney Disease, Effects of kidney disease on your daily life and Satisfaction with treatment. The scores on each dimension range from 0 (worst) to 100 range (better).
Depression, anxiety and stress | Change from Baseline in DASS-21 at 6 months
  The Depression, Anxiety and Stress Scale DASS-21 is a self-report scale containing three subscales scored in a four-point Likert format, ranging from 0 ("Strongly Disagree") to 3 ("Strongly Agree") in increasing order of symptom severity and frequency. Each subscale of the DASS consists of seven items that assess the states of depression (range 0-21), anxiety (range 0-20) and stress (range 0-21), where higher scores are indicative of higher levels of psychological distress.
Interest in Mindfulness | Change from Baseline in Interest in Mindfulness at 6 months
  Analogue scale of interest in mindfulness where participants must fill in a scale of 1 to 10, how much they are interested in mindfulness practices, where 1 corresponds to "I am not at all interested" and 10 corresponds to "I am very interested".
Level of Mindfulness | Change from Baseline in FFMQ at 6 months
  The Five Facet Mindfulness Questionnaire (FFMQ) is a self-report scale that measures the level of Mindfulness through a multidimensional evaluation of its five facets: non-reactivity to inner experience, observe, act with awareness, describe and not judgment of inner experience. It includes 39-items that are rated on a 5-point Likert-type scale ranging from 1 (never or very rarely true) to 5 (very often or always true), with higher scores indicating higher levels of mindfulness skills.
Pain Profile | Change from Baseline in PCP:S at 6 months
  The Profile of Chronic Pain: Screen (PCP:S) is a self-report scale with fifteen items that allow the rapid identification of the pain experience on a multidimensional level of an individual. It is divided into three dimensions: frequency and intensity of pain (four items; score from 0 to 30), interference of pain in daily activities (six items; score from 0 to 36) and effect of pain on emotions (five items; score from 0 to 25). It guides patients to assess the frequency of any pain, average pain, severity, and the highest pain intensity over the past 6 months.
Self-Compassion | Change from Baseline in SCS at 6 months
  The Self-Compassion Scale (SCS) is a self-report questionnaire that includes three basic components: self kindness (extend gentleness and understanding to self rather than self-criticism), ordinary humanity (see your experience as a part of the human experience, rather than being isolated) and Mindfulness (not over-identification with thoughts and more painful feelings). The answers are given on a likert scale (1- "almost never" to 5 "almost always"), when the answers are not compassionate they must be calculated inversely.
Biological markers | Change from Baseline in C-reactive protein and interleukin 6 at 6 months
  Plasma concentrations of inflammatory markers (C-reactive protein and interleukin 6) will be measured.
Inquiry of the Mindfulness Practice | During the 8 weeks of Intervention
  In each mindfulness session, after the practices, an inquiry will be carried out focused on the participant's described experience, where one describes bodily sensations, emotions and thoughts perceived during the practice. This description is made from the investigation of the mindfulness instructor.
Interviews | During the 8 weeks of Intervention and after intervention
  Interviews will be carried out with participants of the studied phenomenon or with key informants who know about the phenomenon or context researched. Conducted individually and semi-structured based on a script designed to ensure coverage of the investigated indicators.
Feasibility of the Hemomindful Program | During the 8 weeks of Intervention and after intervention
  Retention to the study protocol will be assessed using the primary data of all participants at the beginning of the study.
  The adherence to the Hemomindful Program, implementation, security, and satisfaction of the treatment will be assessed through all the participants of the Intervention Group.

CONTACTS AND LOCATIONS:
Overall Officials: Angélica N Adamoli, MD, Principal Investigator — Nephrology Service Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil